CLINICAL TRIAL: NCT00026442
Title: A Pilot Trial Of Two Different Doses Of Capecitabine (XELODA) In Patients With Advanced And/Or Metastatic Breast Cancer
Brief Title: Capecitabine in Treating Women With Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Pharmatech Oncology (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000069030; PHARMATECH-XEL-154; PHARMATECH-20010330; ROCHE-PHARMATECH-XEL-154
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2004-04

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to compare the effectiveness of two different doses of capecitabine in treating women who have advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the objective response rate in women with advanced or metastatic breast cancer treated with two dose levels of capecitabine.
* Compare the duration of response, time to progression, time to treatment failure, survival, incidence of adverse events, and time to onset of the adverse experience in patients treated with this drug.
* Compare the quality of life of patients treated with this drug.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to Karnofsky performance status (70-80% vs 90-100%) and presence of hepatic metastases (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive lower-dose oral capecitabine twice daily on days 1-14.
* Arm II: Patients receive higher-dose oral capecitabine twice daily on days 1-14.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at the end of the third and sixth courses, and at completion of therapy.

PROJECTED ACCRUAL: A total of 120 patients (60 per treatment arm) will be accrued for this study within 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and/or cytologically confirmed breast cancer
* Advanced and/or metastatic disease
* At least 1 measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No CNS metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase no greater than 2.5 times ULN (5 times ULN if liver metastases present OR 10 times ULN if bone metastases present)
* No hepatitis

Renal:

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No clinically significant cardiac disease
* No congestive heart failure
* No symptomatic coronary artery disease
* No cardiac arrhythmias poorly controlled with medication
* No myocardial infarction within the past 12 months even if adequately controlled with medication

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No severe pain inadequately controlled by analgesics
* No prior severe and unexpected reaction to fluoropyrimidine therapy
* No known hypersensitivity to fluorouracil
* No impaired physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome
* No inability to swallow tablets
* No history of uncontrolled seizures, central nervous system disorder, or psychiatric disability that would preclude study participation
* No serious uncontrolled infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 2 but no more than 3 prior chemotherapy regimens
* At least 1 prior chemotherapy regimen containing paclitaxel and an anthracycline as adjuvant therapy or for advanced and/or metastatic disease

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to target lesions unless there is evidence of new disease within the irradiated field
* No concurrent radiotherapy

Surgery:

* No prior organ allografts

Other:

* At least 4 weeks since prior investigational drug
* No concurrent enrollment on other investigational study
* No other concurrent anticancer agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11

CONTACTS AND LOCATIONS:
Overall Officials: Sandy Marcus, Study Chair — Pharmatech Oncology
Locations (10):
- United States (10):
  - Antelope Valley Hospital, Lancaster, California
  - Medical Oncology Care Associates, Orange, California
  - California Cancer Medical Center, West Covina, California
  - Oncology Clinic, P.C., Colorado Springs, Colorado
  - Hematology Oncology Associates of theTreasure Coast - Port St. Lucie, Port Saint Lucie, Florida
  - North Florida Cancer Center, Saint Augustine, Florida
  - Maryland Hematology/Oncology Associates, Baltimore, Maryland
  - Charleston Hematology-Oncology, P.A., Charleston, South Carolina
  - Family Cancer Center, Collierville, Tennessee
  - Logan Regional Hospital, Logan, Utah